CLINICAL TRIAL: NCT06980246
Title: Clinical Utility of Upper-extremity Plyometrics for Enhancing Muscle Strength and Functional Capabilities in Children With Hemiparetic Cerebral Palsy: a Randomized Controlled Trial
Brief Title: Utility of Upper-Extremity Plyometrics in Children With Unilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0023/0013
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: A prospective, two-arm, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blind to the allocation of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyo-Ex group (Experimental): Children in this group received the Plyo-Ex program
  Interventions: Other: Plyometric Exercise
- Control group (Active Comparator): Children in this group received the standard exercise program.
  Interventions: Other: Standard exercise program

INTERVENTIONS:
Other: Plyometric Exercise — The Plyo-Ex program was conducted for 45 minutes/session twice weekly over 12 weeks. The program was directed by a pediatric physical therapist in accordance with the safety performance guidelines defined by the American Academy of Pediatrics and the US National Strength and Conditioning Association. The program consisted of ten unilateral and bilateral upper extremity exercises in the form of push-ups and ball slams/throws/passes activities and was preceded by a warm-up for 5 minutes and ended with a cool-down for 5 minutes.
  Arms: Plyo-Ex group
Other: Standard exercise program — The standard exercise program lasted for 45 minutes/session and repeated two times a week for 12 consecutive weeks. The program was conducted by a pediatric physical therapist and consisted of flexibility exercises, strength training, weight-bearing exercises, proprioceptive neuromuscular facilitation, coordination exercise, and functional training.
  Arms: Control group

SUMMARY:
This study was set out to evaluate the effect of a 12-week upper extremity plyometric exercise (Plyo-Ex) on muscle strength and upper extremity function in children with hemiparetic cerebral palsy (Hemi-CP). Fifty-eight children with Hemi-CP were randomly allocated to the Plyo-Ex group (n = 29, received Plyo-Ex program, twice/week, over 12 weeks) or the control group (n = 29, received standard exercise program). Both groups were assessed for muscle strength and upper extremity function before and after treatment.

DETAILED DESCRIPTION:
Fifty-eight children with Hemi-CP were recruited from the Physical Therapy Outpatient Clinic of Prince Sattam Bin Abdulaziz University and three referral hospitals in Riyadh provenience, Saudi Arabia. Their age ranged between 10 and 15 years, were functioning at levels I or II according to the Gross Motor Function Classification System, and had spasticity levels 1 or 1+ per the Modified Ashworth Scale. Children were excluded if they had fixed deformities, underwent neuromuscular or orthopedic surgery in the last 12 months, submitted to BOTOX injection in the past 6 months, had attentional neglect, demonstrated any cognitive issues, and if they had cardiopulmonary problems that could be exacerbated by exercise.

Outcome measures

Muscle strength: The peak isometric muscle strength of the shoulder flexors, abductors, external rotators, elbow extensors, and wrist extensors was measured using a hand-held dynamometer.

Unilateral upper-extremity function : The unimanual functional performance was assessed using Melbourne Assessment (MA).

Bimanual hand function:The biimanual functional performance was evaluated utilizing the Assisting Hand Assessment (AHA)

The Plyo-Ex group received a 12-week therapist-led Plyo-Ex training, for approximately 45 minutes per session, two times a week for 12 consecutive weeks, in conformity with the National Strength and Conditioning Association guidelines and American Academy of Pediatrics safety standards. The Plyo-Ex program consisted of ten unilateral and bilateral upper extremity exercises in the form of push-ups and ball slams/throws/passes activities. The Plyo-Ex program preceded with a warm-up for 5 minutes and ended with a cool-down for 5 minutes. The control group received the standard exercise program, 45 minutes per session, two times a week for 12 consecutive weeks. The program consisted of flexibility exercises, strength training, weight-bearing exercises, proprioceptive neuromuscular facilitation, coordination exercise, task-oriented training, and functional exercises.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral cerebral palsy
* Age 10-15 years
* Motor function level I or II according to the Gross Motor Function Classification System.
* Spasticity level 1 or 1+ according to the Modified Ashworth Scale

Exclusion Criteria:

* Structural deformities/contractures
* Musculoskeletal or neural surgery in the last year
* BOTOX injection in the last 6 months.
* Cardiopulmonary disorders that could be exacerbated by exercise.
* Perceptual and/or behavioral disorders.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2023-02-12 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 2 months
  The peak isometric muscle strength (Kg) was measured using a hand-held dynamometer

SECONDARY OUTCOMES:
Unilateral upper-extremity function | 2 months
  The unilateral upper-extremity function was assessed using the Melbourne Assessment (MA), which includes 16 standardized tasks assessing reaching, grasping, releasing, and manipulation. It was administered with the child seated at a table, and sessions were video recorded for later scoring. Each task is scored on a 3-5-point scale based on movement quality, accuracy, fluency, dexterity, and speed, yielding 37 sub-scores. Total scores (max 122) are converted to a percentage; higher values indicate better function.
Spontaneity of the upper extremity use | 2 months
  Spontaneity of upper extremity use was assessed using the Shriners Hospital Upper Extremity Evaluation (SHUEE), a video-based tool that evaluates spontaneous movement of the elbow, forearm, wrist, thumb, and fingers during 9 out of 16 standardized tasks. The Spontaneous Functional Analysis (SFA) score is rated on a 6-point scale (0 = no use, 5 = optimal use), with a maximum score of 45 indicating normal spontaneous function.
Dynamic positional alignment of the upper extremity | 2 months
  The dynamic positional alignment (DPA) of the upper extremity was evaluated using the Shriners Hospital Upper Extremity Evaluation (SHUEE), a video-based assessment that examines the alignment of five segments (thumb, fingers, wrist, forearm, elbow) during 16 standardized tasks. For DPA, each segment is scored across four tasks using a 4-point scale (0 = poor alignment, 3 = normal alignment). Total DPA score is the sum of all segment scores, with a maximum of 72 indicating optimal alignment.
Grasp-release Ability | 2 months
  The grasp-release ability (GRA) was assessed using the Shriners Hospital Upper Extremity Evaluation (SHUEE), a video-based tool that evaluates the ability to grasp and release objects with the wrist in flexion, neutral, and extended positions. Each trial is scored on a binary scale (0 = cannot perform, 1 = can perform), with a maximum score of 6 indicating normal or optimal function
Bimanual hand function | 2 months
  The bimanual hand function was assessed using the Assisting Hand Assessment (AHA), a standardized tool for children and adolescents (18 months to 18 years) with unilateral disabilities. It evaluates use of the affected hand during 22 bimanual tasks, scored on a 4-point scale. Raw scores range from 22 to 88, with higher scores indicating better performance. Results were converted to logit-based AHA units (0-100) and reported as such.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elnaggar RK, Ramirez-Campillo R, Elfakharany MS, Alrawaili SM, Alghadier M, Alotaibi MA, El-Basatiny HM, Elsaeed TM. Task-Oriented Plyometric Intervention for Augmenting Upper Extremity Strength and Function in Hemiparetic Cerebral Palsy: A Randomized Controlled Trial. NeuroRehabilitation. 2025 Dec 24:10538135251400762. doi: 10.1177/10538135251400762. Online ahead of print. PMID 41442215